CLINICAL TRIAL: NCT05072717
Title: Single-center Pilot Prospective Observational Study to Determine Feasibility of Assessing Meniscal Tissue Vascularity Using Dynamic Contrast-enhanced Fluorescence Arthroscopy
Brief Title: Dynamic Contrast-Enhanced Fluorescence Arthroscopy of Meniscus Pilot
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: At the time of writing the protocol, was unaware that there is already an established protocol in place within Geriatrics department to capture this data.
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: KARL STORZ Endoscopy-America, Inc. (Industry)
Responsible Party: Principal Investigator, Michael B. Sparks, Associate Professor of Orthopaedics, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY02000782
Record Dates: First submitted 2021-09-09; First posted 2021-10-11 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Knee Injuries
Keywords: meniscus; Indocyanine green; fluorescence; imaging
MeSH Terms: conditions — Knee Injuries | interventions — Perfusion; Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with a meniscal tear requiring surgery (Experimental): Patients will be administered Food and Drug Administration (FDA) approved Indocyanine green (ICG) through intravenous injection and imaged by a FDA approved surgical fluorescence imaging device. Both ICG fluorescence and the imaging system have been used for routine clinical practice for many years. ICG fluorescence imaging utilizes intravenously injected ICG, which is a fluorescent dye that is FDA-approved for clinical use, illuminated with near-infrared light. The ICG dye is indirectly activated and the dynamic fluorescence due to meniscal perfusion can be captured by an arthroscopic imaging system.
  Interventions: Procedure: Perfusion with Indocyanine green

INTERVENTIONS:
Procedure: Perfusion with Indocyanine green — Infusion of Indocyanine green to determine perfusion in meniscal tear tissue.

SUMMARY:
Single-center pilot prospective observational study to determine feasibility of assessing meniscal tissue vascularity using dynamic contrast-enhanced fluorescence arthroscopy

DETAILED DESCRIPTION:
The purpose of this pilot study is to determine whether it is possible to translate the dynamic contrast-enhanced fluorescence imaging methods we have been using to assess bone perfusion in orthopaedic trauma patients to the field of arthroscopic surgery. In other words, it is the development of dynamic contrast-enhanced fluorescence arthroscopy.

While fluorescence arthroscopes are available, there are several challenges associated with minimally invasive procedures compared with wide field imaging, and this pilot study will help determine whether these can be overcome. They are mainly to do with motion artifacts caused by the non-fixed position of the scope during wash-in/wash-out of the dye, and the use of an arthroscopic pump to pressurize the fluid in the surgical cavity.

The long-term goal of this work is to use dynamic contrast-enhanced fluorescence arthroscopy for the assessment of vascularity of meniscal tissue arthroscopically to determine potential healing capacity using dynamic contrast-enhanced fluorescence imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older.
2. Meniscal tear based on MRI or preoperative assessment
3. Provision of informed consent.

Exclusion Criteria:

1. Inability of patient to provide informed consent
2. Iodine allergy.
3. Evidence of septic arthritis of the proposed surgical joint.
4. Burns.
5. Incarceration.
6. Expected survival of less than 90 days.
7. Problems, in the judgment of study personnel, with maintaining follow-up with the patient.
8. Pregnant or Breastfeeding Women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of meniscal blood supply using Indocyanine green (ICG) | Baseline, up to 20 minutes
  The primary study outcome is to measure meniscal blood flow in patients during surgery.

SECONDARY OUTCOMES:
Pressure setting (mm Hg) required for optimal visualization of ICG-based fluorescence. | Baseline, up to 20 minutes
  assess the impact of arthroscopic pump pressure on the visualization of ICG-based dynamic contrast-enhanced fluorescence in the joint and to develop parameters around effect of the pump.

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Sparks, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liao D, Xie L, Han Y, Du S, Wang H, Zeng C, Li Y. Dynamic contrast-enhanced magnetic resonance imaging for differentiating osteomyelitis from acute neuropathic arthropathy in the complicated diabetic foot. Skeletal Radiol. 2018 Oct;47(10):1337-1347. doi: 10.1007/s00256-018-2942-4. Epub 2018 Apr 13. PMID 29654348
- [Background] Fischer C, Nissen M, Schmidmaier G, Bruckner T, Kauczor HU, Weber MA. Dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) for the prediction of non-union consolidation. Injury. 2017 Feb;48(2):357-363. doi: 10.1016/j.injury.2017.01.021. Epub 2017 Jan 9. PMID 28088373
- [Background] Fischer C, Preuss EM, Tanner M, Bruckner T, Krix M, Amarteifio E, Miska M, Moghaddam-Alvandi A, Schmidmaier G, Weber MA. Dynamic Contrast-Enhanced Sonography and Dynamic Contrast-Enhanced Magnetic Resonance Imaging for Preoperative Diagnosis of Infected Nonunions. J Ultrasound Med. 2016 May;35(5):933-42. doi: 10.7863/ultra.15.06107. Epub 2016 Apr 1. PMID 27036169
- [Background] Muller G, Mansson S, Muller MF, Johansson M, Bjorkman A. Increased perfusion in dynamic gadolinium-enhanced MRI correlates with areas of bone repair and of bone necrosis in patients with Kienbock's disease. J Magn Reson Imaging. 2019 Aug;50(2):481-489. doi: 10.1002/jmri.26573. Epub 2018 Dec 16. PMID 30556360
- [Background] Schoierer O, Bloess K, Bender D, Burkholder I, Kauczor HU, Schmidmaier G, Weber MA. Dynamic contrast-enhanced magnetic resonance imaging can assess vascularity within fracture non-unions and predicts good outcome. Eur Radiol. 2014 Feb;24(2):449-59. doi: 10.1007/s00330-013-3043-3. Epub 2013 Oct 22. PMID 24145951
- [Background] Martin Noguerol T, Luna Alcala A, Beltran LS, Gomez Cabrera M, Broncano Cabrero J, Vilanova JC. Advanced MR Imaging Techniques for Differentiation of Neuropathic Arthropathy and Osteomyelitis in the Diabetic Foot. Radiographics. 2017 Jul-Aug;37(4):1161-1180. doi: 10.1148/rg.2017160101. PMID 28696850
- [Background] Cahill RA, Ris F, Mortensen NJ. Near-infrared laparoscopy for real-time intra-operative arterial and lymphatic perfusion imaging. Colorectal Dis. 2011 Nov;13 Suppl 7:12-7. doi: 10.1111/j.1463-1318.2011.02772.x. PMID 22098511
- [Background] Reinhart MB, Huntington CR, Blair LJ, Heniford BT, Augenstein VA. Indocyanine Green: Historical Context, Current Applications, and Future Considerations. Surg Innov. 2016 Apr;23(2):166-75. doi: 10.1177/1553350615604053. Epub 2015 Sep 10. PMID 26359355
- [Background] Valerio I, Green JM 3rd, Sacks JM, Thomas S, Sabino J, Acarturk TO. Vascularized osseous flaps and assessing their bipartate perfusion pattern via intraoperative fluorescence angiography. J Reconstr Microsurg. 2015 Jan;31(1):45-53. doi: 10.1055/s-0034-1383821. Epub 2014 Dec 3. PMID 25469765
- [Background] Alander JT, Kaartinen I, Laakso A, Patila T, Spillmann T, Tuchin VV, Venermo M, Valisuo P. A review of indocyanine green fluorescent imaging in surgery. Int J Biomed Imaging. 2012;2012:940585. doi: 10.1155/2012/940585. Epub 2012 Apr 22. PMID 22577366
- [Background] Boni L, David G, Mangano A, Dionigi G, Rausei S, Spampatti S, Cassinotti E, Fingerhut A. Clinical applications of indocyanine green (ICG) enhanced fluorescence in laparoscopic surgery. Surg Endosc. 2015 Jul;29(7):2046-55. doi: 10.1007/s00464-014-3895-x. Epub 2014 Oct 11. PMID 25303914